CLINICAL TRIAL: NCT07330778
Title: An Open-Label, Single-Dose Study to Assess the Safety, Pharmacodynamics, and Pharmacokinetics of CDX-622 in Adults With Mild to Moderate Asthma
Brief Title: A Study of CDX-622 in Participants With Mild to Moderate Asthma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX622-02
Record Dates: First submitted 2025-09-26; First posted 2026-01-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mild to Moderate Asthma
Keywords: Asthma; Mild to moderate; CDX-622
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-622 (Experimental): Eligible participants will receive a single dose
  Interventions: Drug: CDX-622

INTERVENTIONS:
Drug: CDX-622 — Administered Intravenously

SUMMARY:
This is a study to determine the safety, pharmacodynamics (PD), and pharmacokinetics (PK) of CDX-622 in adults with mild to moderate asthma.

DETAILED DESCRIPTION:
CDX-622 is a bispecific antibody that binds to stem cell factor (SCF) and thymic stromal lymphopoietin (TSLP). Eligible participants with mild to moderate asthma will receive a single dose of CDX-622 via IV infusion. Additional follow-up visits will be required through EOS (week 12).

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, ≥ 18 years of age
2. Diagnosis of mild to moderate asthma for at least 12 months
3. Pre-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 70% of predicted normal
4. Airway reversibility ≥ 12% and 200 mL improvement in FEV1
5. Both males and females of child-bearing potential must agree to use contraception during the study and for 150 days after treatment
6. Willing and able to comply with all study requirements and procedures

Key Exclusion Criteria:

1. Females who are pregnant or nursing
2. Pulmonary disease other than asthma
3. Systemic diseases with elevated eosinophils other than asthma
4. Hospitalization or oral corticosteroids due to asthma within the past 6 months
5. History of needing ventilator support due to asthma
6. Current nasal polyps
7. Severe or uncontrolled asthma
8. History of smoking or vaping within the past 12 months
9. Tuberculosis, hepatitis B or C virus, or HIV
10. Immunomodulating biologic therapies within the past 3 months
11. Prior receipt of TSLP or KIT inhibitors such as tezepelumab or briquilimab

Additional protocol defined inclusion and exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability profile of CDX-622 in adults with mild to moderate asthma. | Day 1 up to Day 85 (12 weeks)
  Occurrence and incidence of Treatment-Emergent Adverse Events (TEAE) and serious adverse events during the study.

SECONDARY OUTCOMES:
Change from baseline in fractional exhaled nitric oxide (FeNO) through week 12. | Day 1 up to Day 85 (12 weeks)
  Pre-treatment and post-treatment FeNO levels will be measured at specified visits and analyzed to evaluate changes from baseline in airway inflammation.
Change from baseline in absolute eosinophil count (AEC) through week 12. | Day 1 up to Day 85 (12 weeks)
  Pre-treatment and post treatment blood samples will be collected at specified visits and analyzed for changes in AEC.
Change from baseline through week 12 in serum biomarkers. | Day 1 up to Day 85 (12 weeks)
  Pre-treatment and post-treatment blood samples will be collected at specified visits and analyzed for changes in TSLP- and SCF-related serum biomarkers.
Pharmacokinetic (PK) evaluation from baseline through week 12. | Day 1 up to Day 85 (12 weeks)
  CDX-622 serum concentrations measured at specific visits.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided